CLINICAL TRIAL: NCT02267785
Title: Exercise Targeting Cognitive Impairment in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern California (Other)
Collaborators: National Parkinson Foundation (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Giselle Petzinger, Assistant Professor of Neurology, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-14-00422
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Parkinson's Disease
Keywords: exercise; mild cognitive impairment; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Skill-Based Exercise (Experimental): Participants assigned to this arm will complete the Skill-Based Exercise Intervention
  Interventions: Other: Skill-Based Exercise
- Aerobic Exercise (Experimental): Participants assigned to this arm will complete the Aerobic Exercise Intervention
  Interventions: Other: Aerobic Exercise
- Social Contact Group (Experimental): Participants assigned to this arm will complete the Social Contact Intervention
  Interventions: Other: Social Contact

INTERVENTIONS:
Other: Skill-Based Exercise — The skill-based exercise program is designed to improve skilled function, fine and gross- motor body coordination. The intervention will be focused on acquisition and improvement of complex movements for the whole body and include the following general categories of activities: (1) balance, (2) eye-hand coordination, (3) leg-arm coordination; 4) reaction time to moving objects/persons; (5) dynamic gait and 6) functional activity performance. The treating therapist will direct both general principles of progression and progression specific to each category.
  Arms: Skill-Based Exercise
Other: Aerobic Exercise — The aerobic cardiovascular exercise will consist of 36 1-hour sessions performed 3 times weekly over 12 weeks. Aerobic exercise will consist of cycling on a recumbent stationary bicycle. Each session will begin and end with gentle stretching. Continuous cycling will be performed for 45-50 minutes, with the first and last 5 minutes designated as warm-up and cool-down periods. The intensity of the middle 30 minutes of cycling will be increased progressively from an initial target of 50% maximum heart rate (HR) during week 1 to 75% of maximum HR by week 12. The initial intensity will be set at 50% of maximum HR. Participants will be encouraged to cycle as fast as they can, with a goal of maintaining 90 revolutions per minute (RPM) throughout the middle 30-minute period. Pedaling resistance will be kept low throughout all sessions. Measures of heart rate via heart rate monitors, blood pressure, RPM, and rate of perceived exertion will be recorded at 5-minute intervals.
  Arms: Aerobic Exercise
Other: Social Contact — The control Social Contact group will consist of an equal amount of social contact as the exercise group. Subjects will have weekly visits at the University of Southern California with the study coordinator. The goal is for 3 hours of social contact every week for a total of 36 hours over 12 weeks. Activities scheduled for the social contact visits will include: (1) support group interactions and (2) social outings such as a trip to a museum, local café for lunch or dinner; (3) book club; (4) sports event. Support group interaction can include discussions among patients and caregivers, presentations from experts in various aspects of PD. They will be instructed to continue with their usual level of activity but refrain from beginning new exercise activities during the study period.
  Arms: Social Contact Group

SUMMARY:
The aim of this application is to compare and elucidate the effects of skill-based versus aerobic exercise versus control on mild cognitive impairment (MCI) of the executive function (EF) subtype in Parkinson's disease (PD); we hypothesize that skill-based exercise will result in the greatest improvement in EF and lead to modification of underlying neural substrates.

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI), particularly of the executive function (EF) subtype, is common in Parkinson's disease (PD) and transitions to dementia, increased fall risk, and poor quality of life. EF is a set of processes that include mental flexibility and attention that are needed to learn and optimize performance of complex cognitive and motor skills. Such skills include the ability to generalize task performance under different conditions (context processing) and to perform two tasks simultaneously termed dual-task (DT) performance. Deficits in EF lead to problems in daily functioning and loss of independence and create psychosocial and economic burdens on patients and caregivers and stakeholders including health care providers. There is currently no effective treatment in PD to address EF deficits. Our animal and clinical studies in PD demonstrate that skilled exercise facilitates neuroplasticity of the basal ganglia (BG), a brain region sub-serving EF and supports the hypothesis that exercise will reverse EF deficits in PD. Furthermore, recent studies in healthy aging support that skill-based exercise that specifically promotes motor skill fitness (MSF), compared with aerobic exercise that promotes cardiovascular fitness (CF), has a greater impact on EF and related BG circuits. The aim of this application is to compare and elucidate the effects of skill-based versus aerobic exercise versus control on MCI of the EF subtype in PD; we hypothesize that skill-based exercise will result in the greatest improvement in EF and lead to modification of underlying neural substrates.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to provide informed consent
* confirmed diagnosis of idiopathic PD based on the United Kingdom Brain Bank criteria
* Mild cognitive impairment (Level II criteria Movement Disorder Task Force)
* medically eligible for MRI imaging
* able to provide a written medical clearance from their primary physician to participate in exercise
* stable PD medications for 3 months

Exclusion Criteria:

* a Hoehn & Yahr staging greater than 2.5 at screening
* severe cardiac disease (New York Heart Association classification IIIV)
* history of an abnormal stress test
* clinically significant medical or psychiatric illness
* electrically, magnetically, or mechanically activated implant (such as cardiac pacemakers or intracerebral vascular clip)
* metal in any part of the body including metal injury to the eye
* past history of brain lesions (such as stroke)
* seizures or unexplained spells of loss of consciousness
* family history of epilepsy
* physical therapy within 6 months of the study
* symptomatic orthostatic hypotension at the screening visit
* orthopedic and other movement-influencing diseases such as arthritis or total hip joint replacement
* requirement for central nervous system active therapies (e.g. hypnotics, antidepressants, anxiolytics)
* moderate or severe depression or apathy using the Geriatric depression scale and Apathy scale
* taking anticholinesterase inhibitors
* taking anticholinergic medication
* PD dementia
* Colorblindness

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in Context Dependent Motor Learning (CDML) | at Baseline, after 12 week intervention, and at 12 week follow up visit
  All subjects from each group will undergo a finger sequence motor learning task to determine exercise effects on EF as evaluated through improvement in the transfer of a learned motor task from one contextual setting to another.
Change in Dual Task Performance and Functional Magnetic Resonance Imaging (fMRI) | at Baseline, after 12 week intervention
  A subset of subjects (60 representing 20 per group) will be invited to undergo fMRI studies at University of California, Los Angeles. Patients will perform a learned single finger-sequencing task (a condition of the CDML) with an additional secondary dual task (DT) component during an fMRI scan.
Change in D-KEFS Verbal Fluency Test | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The D-KEFS Verbal Fluency test will be used to evaluate executive function
Change in Tower of London Test | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The Tower of London test will be used to evaluate executive function
Change in Wisconsin Card Sorting Test | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The Wisconsin Card Sorting test will be used to evaluate executive function

SECONDARY OUTCOMES:
Change in Parkinson Disease Questionnaire-39 (PDQ-39) | at Baseline, after 12 week intervention, and at 12 week follow up visit
  Parkinson Disease Questionnaire-39 (PDQ-39) will be used to indicate overall quality of life and frequency with which patients experience difficulties; high scores for the PDQ-39 reflect poorer quality of life.
Change in Evaluation of PD Motor Symptoms with Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The MDS-UPDRS is the established gold standard that is currently used for the vast majority of clinical settings and for scientific trials. This scale was developed in 1987 and is the most widely used tool in PD.
Change in Activity Specific Balance Confidence (ABC) Scale | at Baseline, after 12 week intervention, and at 12 week follow up visit
  Activity Specific Balance Confidence (ABC) Scale is a 16-item self-report in which patients rate their balance confidence in performing several activities; high scores indicate greater balance confidence.
Change in Confidence in ability to maintain an exercise program (CONF) | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The CONF scale includes nine items, which assesses how sure subjects are that they would do exercise under different conditions or constraints, including when they are tired.
Change in Exercise Control Beliefs (BEL) | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The BEL, 6-item scale was developed to assess beliefs about control over exercise behavior.
Change in Self-efficacy for Exercise Scale (EFFIC) | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The EFFIC scale is a self-efficacy barriers to exercise measure, a 13-item instrument that focuses on self-efficacy expectations related to the ability to continue exercising in the face of barriers to exercise.
Change in Frontal Systems Behavior Scale (FrSBe) | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The FrSBe assesses changes in behavior dysfunction and disturbances associated with frontal-subcortical damage, which is the circuitry involved with executive functioning
Change in Motor Skill Fitness | at Baseline, after 12 week intervention, and at 12 week follow up visit
  An individual's Motor skill fitness will be a composite score of their Physical Performance Test (PPT) and their Timed Up and Go (TUG).
Change in Cardiovascular Fitness | at Baseline, after 12 week intervention, and at 12 week follow up visit
  Subjects will participate in testing designed to determine their level of cardiovascular fitness by estimating maximal oxygen uptake (V02max) known as the Balke treadmill submaximal fitness test and has been optimized for use in samples of elderly adults.
Change in Lifetime Total Physical Activity Questionnaire (LTPAQ) | at Baseline
  The LPAQ measures the time spent in physical activity over the lifetime of the subject
Change in Global Physical Activity Questionnaire (GPAQ) | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The GPAQ measures the time spent in physical activity during a normal week
Change in Body Mass Index | at Baseline, after 12 week intervention, and at 12 week follow up visit
Change in Body Fat Percentage | at Baseline, after 12 week intervention, and at 12 week follow up visit
Change in Mattis Dementia Rating Scale | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The Mattis Dementia Rating Scale will be used to differentiate between study subjects with mild cognitive impairment and dementia
Change in Geriatric Depression Scale | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The Geriatric Depression Scale will be used to evaluate study subjects for depression
Change in Geriatric Anxiety Inventory | at Baseline, after 12 week intervention, and at 12 week follow up visit
Change in Apathy Scale | at Baseline, after 12 week intervention, and at 12 week follow up visit
Change in Revised Activities of Daily Living Scale | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The Revised Activities of Daily Living Scale will be used to evaluate independent living skills
Change in the Frontal Systems Behavior Scale (FrSBe) | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The FrSBe will be used to evaluate frontal systems behavior
Change in Adaptive Digit Ordering Test | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The Adaptive Digit Ordering Test will be used to evaluate attention and working memory
Change in Hooper Visual Organization Test | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The Hooper Visual Organization Test will be used to evaluate visuospatial function
Change in Benton's Judgment of Line Orientation | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The Benton's Judgment of Line Orientation test will be used to evaluate visuospatial function
Change in D-KEFS Color Word Interference Test | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The D-KEFS Color Word Interference Test will be used to evaluate attention, working memory and executive function
Change in California Verbal Learning Test- 2nd Edition (CVLT-II) | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The CVLT-II will be used to evaluate memory function
Change in WMS-II Visual Reproduction Test | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The WMS-II Visual Reproduction Test will be used to evaluate memory function
Change in WAIS-IV Similarities Test | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The WAIS-IV Similarities test will be used to evaluate language function
Change in Boston Naming Test | at Baseline, after 12 week intervention, and at 12 week follow up visit
  The Boston Naming Test will be used to evaluate language function

CONTACTS AND LOCATIONS:
Overall Officials: Giselle M Petzinger, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886